CLINICAL TRIAL: NCT04459364
Title: The Prevalence of Pulmonary Hypertension, With or Without Right Ventricular Loading, in Patients With COVID-19 Who Are Being Treated With a Respirator in the Intensive Care Unit.
Brief Title: The Prevalence of Pulmonary Hypertension in Patients With COVID-19.
Status: Completed | Type: Observational
Sponsor: Attgeno AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 20200422PA
Record Dates: First submitted 2020-07-03; First posted 2020-07-07 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Hypertension, Pulmonary; Right Ventricular Overload; COVID
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The virus infection Covid-19 fills our hospitals and intensive care departments in a very unique way and there is a lack of essential insight into the pathophysiology of the disease. As a result, very specific treatment options are missing. The US Medicines Agency (FDA) has in the last days given a general license for treatment with inhaled nitric oxide (iNO). Inhaled NO in Sweden (and Europe) is approved for the indication of pulmonary hypertension in adults.

However, no one has yet described the occurrence of pulmonary hypertension, with or without right ventricular loading, in the Covid-19 patients who become so seriously ill that they need to be treated at an IVA ward. Knowledge of this is, of course, a prerequisite for determining the need for pulmonary artery catheterization (PA catheter, Swan-Ganz catheter) and also to better understand whether iNO treatment or other forms of lung selective vasodilation therapy may be of benefit to this patient group.

DETAILED DESCRIPTION:
Demographics and data from study variables will be documented in paper CRFs at the investigational site.

* Demography

  o Age, sex
* Covid-19 related variables

  o COVID-19 diagnosis
* Concomitant diseases

  o Comorbidity, previous and present
* Cardiovascular risk factors

  o Smoking
* Laboratory values
* On-site measurements o Evaluation with echocardiography

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age
* Diagnosed with COVID-19 and is treated at an intensive care unit.

Exclusion Criteria:

* Responsible investigator considers that co-morbidity is so pronounced that it does not allow reasonable interpretation of data.
* Missing verified diagnosis of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a non-interventional retrospective study to be performed in an intensive care unit in Sweden. The study will include 80 Covid-19 patients who had been examined with echocardiography. Data will be collected through chart review.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Prevalence | Day 1
  To determine the prevalence of pulmonary hypertension and right ventricular load in patients with COVID-19 treated in intensive care unit evaluated by routine echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Arne Lönnqvist, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data that underlie the results reported in this article will be shared, after deidentification (text, figures and appendices)
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal and to achieve aims in the proposal. Proposals should be directed to per-arne.lonnqvist@ki.se. To gain access, data requestors will need to sign a data access agreement.